CLINICAL TRIAL: NCT00873210
Title: Non-Interventional Study In Patients With Advanced And/Or Metastatic Renal Cell Carcinoma (mRCC) Treated With Sutent
Brief Title: Study In Patients With Kidney Cancer Treated With Sutent
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181185
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Advanced or Metastatic Renal Cell Carcinoma; Renal Cancer
Keywords: renal cell carcinoma; sunitinib malate
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Sutent: 125 consecutive patients in outpatient care with advanced or metastatic renal cell carcinoma, that are indicated for 1st or 2nd line anticancer therapy
  Interventions: Drug: Sutent

INTERVENTIONS:
Drug: Sutent — 50 mg per day for 4 consecutive weeks, followed by 2 weeks treatment pause
  Other Names: sunitinib malate

SUMMARY:
Objective of this study is to increase knowledge about safety, tolerability, quality of life and efficacy under conditions of routine use of sunitinib.

DETAILED DESCRIPTION:
Consecutive patients with advanced or metastatic renal cell carcinoma, that are indicated for 1st or 2nd line anticancer therapy

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with advanced or metastatic renal cell carcinoma, that are indicated for 1st or 2nd line anticancer therapy

Exclusion Criteria:

* Hypersensitivity to sunitinib malate or to any of the excipients
* Any other contraindication to the use of sunitinib malate (based on decision of the treating physician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic renal cell carcinoma, that are indicated for 1st or 2nd line anticancer therapy.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Increased knowledge about safety, tolerability, quality of life and efficacy under conditions of routine use of sunitinib | 36 months

SECONDARY OUTCOMES:
Dose modifications | 36 months
Incidence of new diagnosed hypertension | 36 months
Incidence of new diagnosed hypothyroidism | 36 months
Safety of sunitinib malate in "real-life" setting | 36 months
Efficacy of sunitinib malate in "real-life" setting | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Slovakia (13):
  - Pfizer Investigational Site, Banská Bystrica
  - Pfizer Investigational Site, Bojnice
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Michalovce
  - Pfizer Investigational Site, Nitra
  - Pfizer Investigational Site, Poprad
  - Pfizer Investigational Site, Prešov
  - Pfizer Investigational Site, Ružomberok
  - Pfizer Investigational Site, Trebišov
  - Pfizer Investigational Site, Trenčín
  - Pfizer Investigational Site, Trnava
  - Pfizer Investigational Site, Žilina

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181185&StudyName=Study%20In%20Patients%20With%20Kidney%20Cancer%20Treated%20With%20Sutent